CLINICAL TRIAL: NCT06401681
Title: Cross-Education Effects of Balance Training in Individuals With Chronic Ankle Instability
Brief Title: Cross-Education for Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Ryan McCann, Associate Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1407520-8
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Balance Training Group; Control Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training (BAL) (Experimental): Within one day of baseline testing, BAL will begin a progressive balance training protocol on the involved limb. The balance training program consists of three 20-minute sessions per week for eight weeks. Post-test assessments for BAL will completed within one week of completing the 8-week training interval.
  Interventions: Other: Balance training
- Control (CON) (No Intervention): After baseline testing, CON will be instructed to continue their normal daily routine. They will not participate in the balance training intervention.

INTERVENTIONS:
Other: Balance training — The balance exercises consist of single limb stances with eyes open and closed, single-leg hops with stabilization, and single-leg hops and reach. Thirty-second breaks will be provided between exercise sets. Progressions for single-leg stance exercises involve longer durations and introduction of unstable surfaces. Progressions for hopping exercises involve longer hopping distances. To progress to the next level, participants must complete a balance training session without any errors. Errors include 1) touching the floor or bracing with the opposite limb, 2) excessive lateral trunk flexion or hip abduction, 3) hands coming off hips (hop tasks) or shoulders (stance tasks), 4) missing the landing target, 5) using the reach leg for a substantial amount of weight bearing.
  Other Names: balance exercise; balance rehabilitation
  Arms: Balance training (BAL)

SUMMARY:
Chronic ankle instability (CAI) results in neuromuscular impairments compromising balance, lumbopelvic stability, and hip strength. Balance training has proven to be an effective intervention for individuals with CAI. Additionally, unilateral balance training for those with CAI has previously led to cross-education effects in which the untrained limb exhibited improved balance performance. However, the ability of unilateral balance training to improve contralateral hip strength and lumbopelvic stability in those with CAI is unknown. The purpose of this study was to determine the cross-education effects of balance training on hip strength and lumbopelvic stability in individuals with CAI.

Thirty individuals with CAI will be randomized into control (CON) and balance (BAL) groups. Baseline testing include a unilateral hip bridge, hip strength, and balance tests of the uninvolved limb. For the unilateral hip bridge, the participant will hold a bridge through the test limb for maximum time. Isometric hip strength will be measured for external rotation (ER), extension (EXT), and abduction (ABD) using a handheld dynamometer. The star excursion balance test (SEBT) requires participants to maintain a single-leg stance while reaching for maximum distance with the opposite leg in three directions: anterior (SEBT-ANT), posterolateral (SEBT-PL), and posteromedial (SEBT-PM). The BAL group will participate in a progressive balance training program three times a week for eight weeks for the involved limb, whereas CON will not. All baseline measures will be reassessed at the end of the 8 weeks. Separate 2-way repeated measures ANOVAs will analyze the effects of group and time on each outcome. Additionally, each group's mean changes from baseline to post-intervention will be assessed with Cohen's d effect sizes. Statistical significance is set a priori at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* All participants were required to have CAI based on guidelines published by the International Ankle Consortium. Participants were required to have a history of at least one acute LAS that resulted in swelling, pain, and at least one day of missed activity. The initial LAS must have occurred at least 12 months before study enrollment and the participants needed to be free of ankle sprains in the past three months. Participants were also required to report at least two events of "giving way" of their ankle, instability, or reinjury within the previous six months. Lastly, participants had to record scores of ≥5 on the Ankle Instability Instrument (AII), >11 on the Identification of Functional Ankle Instability (IdFAI), and <24 on the Cumberland Ankle Instability Tool (CAIT).2 One member of the research team completed all screening procedures. The same person block randomized participants into two groups, control (CON) and balance training (BAL), by selecting a sealed envelope that contained group designation.

Exclusion Criteria:

* Participants were excluded if they had any history of lower extremity or spine fracture or surgery, any lower extremity or spine injury besides LAS within the past two years, and any significant ankle injury within the past three months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test of the Uninvolved Limb | 10 minutes
  The Star Excursion Balance Test (SEBT) measured balance performance through a series of lower body reaches in anterior, posterolateral, and posteromedial directions. Participants maintained a single-leg stance on the uninvolved limb while reaching with their non-stance limb for maximal distance along a tape measure fixed to the floor. Participants were required to maintain their hands on their hips and keep their stance limb flat against the floor. As a common practice, there were four practice trials and three test trials for each direction performed. For each SEBT direction, we averaged the three reach scores and normalized them as a percent of the stance leg length, measured from the anterior superior iliac spine to the most distal part of the medial malleoli.
Isometric hip strength of the Uninvolved Limb | 15 minutes
  Isometric hip strength was measured via handheld dynamometry for extension, abduction, and external rotation. Participants completed one practice trial and three test trials for each motion in random order. Each trial lasted 5 seconds, with the first 3 seconds gradually increasing force and then the final two seconds exerting maximum force. We averaged the three trials for each hip strength test, multiplied by the length of the moment arm, and divided by body mass to calculate normalized torque (Nm/kg). We measured EXT and ABD moment arms from the greater trochanter to the lateral femoral epicondyle and ER moment arm from the medial tibial plateau to the distal end of the medial malleolus.
Lumbopelvic stability of the Uninvolved Limb | 2 minutes
  We measured lumbopelvic stability with a unilateral hip bridge test. Participants began in a hook-lying position with their arms folded across their chest. Participants completed an initial double-leg bridge to find a neutral alignment of the spine and hips.To start the unilateral hip bridge, participants initiated another bilateral hip bridge, then extended the non-test knee and kept their thighs in parallel. Participants completed a single trial for maximal time (s).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCann, PhD, Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University Athletic Training Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No